CLINICAL TRIAL: NCT06586307
Title: Assessment of DNA Methylation Signatures in Lymphocytes for Evaluating the Efficacy and Prognosis of Immunotherapy in Colorectal Cancer
Brief Title: Estimating Lymphocyte Counts from DNA Methylation
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Head of Gastroenterology, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: MeTIL-01
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancers; Immunotherapy; DNA Methylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: quantitative analysis of DNA methylation at single-base resolution (QASM) — qPCR-based quantitative analysis for single-base methylation (QASM) The methylation percentage of each candidate CpG site was determined in multiple cohorts using a MethyLight-based QASM assay that has been developed and validated in our previous work. In short, the bisulfite-converted DNA was amplified, in which we exploited the locus-specific PCR primers flanking a pair of methylated and unmethylated probes labeled with the fluorescent dyes 6-carboxyfluorescein (6-FAM) and 2-chloro-7phenyl-1,4-dichloro-6-carboxyfluorescein (VIC), respectively. The methylation percentage was calculated by methylation/(methylation+unmethylation)×100%. QASM was performed using the Applied Biosystems QuantStudio 7 Flex Real-Time PCR System (Thermo).

SUMMARY:
The goal of this observational study is to assess lymphocyte levels in colorectal cancer patients using DNA methylation levels in tissues or blood. The main questions it aims to answer are:

Can DNA methylation features calculate lymphocyte levels? Can the calculated lymphocyte levels assess the efficacy and prognosis of immunotherapy?

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with colorectal cancer by colonoscopy pathology and deemed eligible for immunotherapy after assessment.
2. Neoadjuvant immunotherapy regimen includes PD-1 or anti-PD-L1.
3. R0 resection is performed after neoadjuvant immunotherapy.
4. Complete immunotherapy efficacy assessment data and follow-up data are available.
5. The tissue bank stores the required whole blood and tissue samples for the experiment.

Exclusion Criteria:

1. Concurrent other malignancies.
2. Neoadjuvant immunotherapy not conducted according to the standard protocol.
3. Severe adverse chemotherapy reactions that lead to the discontinuation of immunotherapy midway.
4. Lack of complete neoadjuvant chemotherapy efficacy assessment data or follow-up data.
5. The tissue bank does not store the required whole blood or tissue samples for the experiment.
6. Patients with concurrent other immune system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we prospectively enrolled 49 patients with advanced-stage CRC who received neoadjuvant immunotherapy as part of their treatment regimens at the Sixth Affiliated Hospital, Sun Yat-sen University from January 2022 to June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | From the date of neoadjuvant therapy until the date when the surgical specimen pathology results are obtained, the duration of neoadjuvant therapy is approximately half a year, with a maximum of one year.
  The complete response rate refers to the percentage of patients who experience a complete disappearance of their disease after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China